CLINICAL TRIAL: NCT07126314
Title: Critical Appraisals at Play: Elevating EM Journal Clubs With Team-Based Competition
Brief Title: Critical Appraisals at Play
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Principal Investigator, Greg Neyman, Principal Investigator, Community Medical Center, Toms River, NJ
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-007
Record Dates: First submitted 2025-07-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Medical Education
Keywords: Emergency Medicine education; Journal club innovation; Gamified learning; Critical appraisal skills; Team-based competition; Resident engagement; Didactic enhancement; Pre/post intervention; Survey-based evaluation; Emergency Medicine residents; Residency training programs

STUDY DESIGN:
Intervention Model Description: Pre and Post Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residency Cohort (Experimental): Full complement of site emergency medicine residents
  Interventions: Other: Competition based Education Format

INTERVENTIONS:
Other: Competition based Education Format — Residents will be organized into 3 teams, each competing to amass points for critiquing articles presented during journal club, for a prize.

SUMMARY:
Pre and Post assessment of knowledge and attitudes on critical appraisal of biomedical literature in Emergency Medicine practice in a cohort of residents with implementation of a competition based educational format.

DETAILED DESCRIPTION:
During the academic year of 2025-2026, the 36 Emergency Medicine residents of a community medicine affiliate of a tertiary medical center will be compete against each other during the journal club didactic. Three residents will be assigned each month, one from each year, to select a journal article matching the curricular content block of that month. Residents will submit their selected article after faculty approval.

Residents will submit their critiques of the journal articles prior to the scheduled journal club via a dedicated residency website. They will focus on potential methodological flaws of the article. This is congruent to how journal club didactics were focused in the past in the institution, so second and third years will have had exposure to this approach.

During journal club, besides having the resident that selected the article briefly present it, resident critiques will be discussed. A single point will be awarded to each resident for each critique they have submitted. For critiques of significant merit, as determined by the faculty, the journal club facilitator will invite the submitting resident to discuss their critique, and will be awarded 2 points. To discourage artificial intelligence (AI) use without learning, critiques will be selected at faculty discretion to be orally explained during journal club to the satisfaction of the faculty. The faculty have determined that if residents utilize AI as a tool to enhance their learning (instead of simply enumerating critiques blindly on a document), this is in service towards the goal of journal club, and should be encouraged.

As a reward, residents that have the highest running score will receive $100 Amazon gift cards, tiered by 1st, 2nd, and 3rd year academic status.

Attitudes towards the importance of critical assessment of scientific literature, self assessments of fluency in scientific literature appraisal, and the effectiveness of journal club, will be conducted via anonymous survey on RedCap at the beginning and end of the academic year. The survey utilized will be the modified version of a previously validated survey used by Haspel2. Additionally, residents will be assigned Journal Club based quizzes from Rosh Review13, a platform tailored for resident education, at the beginning and end of the year. Rosh Review provides comparative benchmarks that can be used to assess resident performance.

ELIGIBILITY:
Inclusion Criteria:

* All emergency medicine residents at study site

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in score in knowledge based quiz | 11 months
  A journal club based quiz, created by Rosh Review, will be administered pre and post. Changes in scores will be noted.

SECONDARY OUTCOMES:
Difference in knowledge quiz compared to benchmark score | 11 months
  Differences in knowledge score compared to benchmark scores Rosh Review maintains
Changes in attitudes regarding comfort in interpreting biomedical literature | 11 months
  Changes in attitudes regarding comfort in interpreting biomedical literature as measured by validated survey
Subjective assessment of value of curriculum | 11 months
  Subjective assessment of value of curriculum by a survey with likert scale and free entry items

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Robert Wood Johnson Barnabas Health Community Medical Center, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLeod RS, MacRae HM, McKenzie ME, Victor JC, Brasel KJ; Evidence Based Reviews in Surgery Steering Committee. A moderated journal club is more effective than an Internet journal club in teaching critical appraisal skills: results of a multicenter randomized controlled trial. J Am Coll Surg. 2010 Dec;211(6):769-76. doi: 10.1016/j.jamcollsurg.2010.08.016. Epub 2010 Oct 29. PMID 21036071
- [Background] Horneff, J, Baldwin, K, Ahn, J.. "The Value of Journal Clubs in Orthopaedic Resident Education." (2010). University of Pennsylvania Orthopedic Journal
- [Background] Dzara K, Frey-Vogel AS. Medical Education Journal Club for the Millennial Resident: An Interactive, No-Prep Approach. Acad Pediatr. 2019 Aug;19(6):603-607. doi: 10.1016/j.acap.2019.05.004. Epub 2019 May 14. PMID 31100347
- [Background] Allon S, Baggett A, Hayes B, Glosemeyer K, Cavo J, Pacha R, Zurko J, Patel N, Kraemer R. Association of a Gamified Journal Club on Internal Medicine Residents' Engagement and Critical Appraisal Skills. J Grad Med Educ. 2023 Aug;15(4):475-480. doi: 10.4300/JGME-D-22-00812.1. PMID 37637345
- [Background] Moharari RS, Rahimi E, Najafi A, Khashayar P, Khajavi MR, Meysamie AP. Teaching critical appraisal and statistics in anesthesia journal club. QJM. 2009 Feb;102(2):139-41. doi: 10.1093/qjmed/hcn131. Epub 2008 Oct 8. PMID 18842683
- [Background] Luc JGY, Fowler CS, Eisenberg SB, Estrera AL, Wolf RK, Choi CW, Lawton JS, Martin LW, Nesbitt JC, Reznik SI, Nguyen TC, Vaporciyan AA, Antonoff MB; Thoracic Education Cooperative Group (TECoG). Multiinstitutional Evaluation of a Debate-Style Journal Club for Cardiothoracic Surgery Trainees. Ann Thorac Surg. 2022 Jul;114(1):327-333. doi: 10.1016/j.athoracsur.2021.07.104. Epub 2021 Sep 20. PMID 34547299
- [Background] Linzer M, Brown JT, Frazier LM, DeLong ER, Siegel WC. Impact of a medical journal club on house-staff reading habits, knowledge, and critical appraisal skills. A randomized control trial. JAMA. 1988 Nov 4;260(17):2537-41. PMID 3050179
- [Background] Wegleitner, Elizabeth and Octavio R Chirino. "Join the Club: Integration of the CREOG Journal Club Curriculum Improves OBGYN Residents Statistical Literacy." Obstetrics & Gynecology (2019): 134():p 48S, October 2019
- [Background] Hartzell JD, Veerappan GR, Posley K, Shumway NM, Durning SJ. Resident run journal club: a model based on the adult learning theory. Med Teach. 2009 Apr;31(4):e156-61. doi: 10.1080/01421590802516723. PMID 19404887
- [Background] Arti Muley, J. Lakhani "Evidence based vs traditional journal clubs: Time to switchover." The Journal of medical research 2015 1(1): 13-17 https://doi.org/10.31254/jmr.2015.1106
- [Background] Haspel RL. Implementation and assessment of a resident curriculum in evidence-based transfusion medicine. Arch Pathol Lab Med. 2010 Jul;134(7):1054-9. doi: 10.5858/2009-0328-OA.1. PMID 20586637
- [Background] Alavi-Moghaddam M, Yazdani S, Mortazavi F, Chichi S, Hosseini-Zijoud SM. Evidence-based Medicine versus the Conventional Approach to Journal Club Sessions: Which One Is More Successful in Teaching Critical Appraisal Skills? Chonnam Med J. 2016 May;52(2):107-11. doi: 10.4068/cmj.2016.52.2.107. Epub 2016 May 20. PMID 27231674